CLINICAL TRIAL: NCT03552640
Title: Accuracy of Digital Three-Dimensional Root Position Prediction Via Digitized Models
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdullah El-Gendi, Dr, Cairo University
Other Study IDs: CEBD-CU-2018-04-19
Record Dates: First submitted 2018-04-25; First posted 2018-06-12 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Orthodontic Appliance Complication
Keywords: Orthodontics; Digitized Models; Root Position

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Measuring the accuracy of a new technique by which root positions can be predicted at the pre-finishing stage of the comprehensive orthoodntic treatment

DETAILED DESCRIPTION:
A CBCT is taken Pre-Treatment

Segmentation of teeth is done from the CBCT exported as STL files and kept aside.

Routine comprehensive orthodontic treatment is done till pre-finishing stage.

Impression for teeth is taken at this timepoint.

A cast is poured and laser scanned.

Now the investigators have segmented teeth and a cast with new crown positions

The investigators will superimpose the teeth on the crowns of the digital cast to obtain the " Predicted Root Position" (PRP)

To check accuracy of this Prediction a CBCT is taken and compared to the prediction to check its accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring orthodontic treatment
* Adult set of permanent dentition
* Non-extraction cases

Exclusion Criteria:

* Syndromic patients

Ages: 12 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients having only permenant teeth and no decidous ones, requiring orthodontic treatment not involving extraction of teeth in their treatment plan
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Root Position Prediction as assessed by Color Map Heat Analysis | 9 months
  Using Color Map Heat Analysis in millimetres

CONTACTS AND LOCATIONS:
Locations (1):
- Orthodontic Department, Cairo, Egypt